CLINICAL TRIAL: NCT06253052
Title: A Pilot Study to Test Benefits of Drinking Clear Fluids Until Called to the Operating Room in Adult Surgical Patients
Brief Title: Benefits of Drinking Clear Fluids Until Called to the Operating Room in Adult Surgical Patients
Acronym: HYDRATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HYDRATE
Record Dates: First submitted 2024-01-05; First posted 2024-02-12 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Anesthesia; Thirst; Due to Deprivation of Water; Aspiration
Keywords: Surgery; Postoperative Nausea and Vomiting; Delirium; Dehydration; Satisfaction, Patient; Headache
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Delirium; Dehydration; Patient Satisfaction; Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (No Intervention): Fasting instructions as given by anaesthesiologist according to national guidelines (6 h solid meal and thick liquids, 2 h clear fluids).
- Instructed guideline adherence (Active Comparator): Patients should not involuntarily fast fluids for longer than 2 h.
  Interventions: Behavioral: Additional pre-OP-visit
- Experimental intervention (Experimental): Patients should not involuntarily fast fluids for longer than 30 min.
  Interventions: Behavioral: Additional pre-OP-visit; Behavioral: Liberal fasting regime

INTERVENTIONS:
Behavioral: Additional pre-OP-visit — OP-schedule is closely monitored and patients will be visited to support and encourage them in drinking clear fluids.
  Arms: Experimental intervention; Instructed guideline adherence
Behavioral: Liberal fasting regime — Patients may drink up to 200 ml clear fluids between 2 h prior to the surgery and the call to operation room.
  Arms: Experimental intervention

SUMMARY:
The purpose of this study is to show if - compared to standard practice - allowing adults undergoing surgical procedures under anaesthesia care to drink clear fluids up to a volume of 200 ml between 2 h prior to the operation and the call to operation room (approximately 30 min prior to anaesthesia induction) will decrease patient thirst and increase patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 18 years)
2. American Society of Anesthesiologists (ASA) physical status classification I-III
3. Undergoing surgical procedure under anaesthesia care: general anaesthesia, regional anaesthesia, combined anaesthesia or monitored anaesthesia care.

The proportion of Patients undergoing general or combined anaesthesia is aimed to exceed 75%

Exclusion Criteria:

1. Absolute indication for rapid sequence induction including but not limited to:

   1. Bowel obstruction including ileus
   2. Stricture and oesophageal disorders including achalasia
   3. Recent polytrauma or trauma of the upper gastrointestinal tract
   4. Acute abdomen/peritonitis including active gastrointestinal bleeding
2. Relative indication for (modified) rapid sequence induction includes, but is not limited to:

   1. Symptomatic gastroesophageal reflux disease, independent of food intake and persistent under medical treatment (PPI)
   2. Hiatus hernia or upside down stomach
   3. Upper gastrointestinal tumour
   4. History of upper gastrointestinal surgery (oesophageal, gastric, duodenum, pancreatic)
   5. Medically confirmed gastroparesis
   6. Severe obesity, defined as body mass index ≥ 40 kg/m2
3. Dysphagia
4. Renal replacement therapy
5. Fluid restriction therapy
6. Pregnancy
7. Expected need for postoperative mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Thirst | Prior to induction of anaesthesia
  At any stage after your hospital admission have you had the following: Thirst (No/ Yes, moderate/ Yes, severe)

SECONDARY OUTCOMES:
Total number of protocol deviations per group | From enrollment until last Follow-up is concluded at up to 48 hours post surgery
  Outcome assessment successfully blinded Real fluid fasting time is less than allocated fluid fasting time
Fluid fasting time | Prior to induction of anesthesia
  Actual fluid fasting time in hours
RASS | 2 hours after end of surgery
  Richmond Agitation Sedation Scale. A scale from -5 to +4 is used. Negative values indicate a sedated state. Positive values indicate an agitated state.
CAM-ICU | 2 hours after end of surgery
  Confusion Assessment Method for the Intensive Care Unit.
Headache | Prior to induction of anesthesia and 2 hours after end of surgery
  At any stage after your hospital admission have you had the following: Headache (No/ Yes, moderate/ Yes, severe)
Change of heart rate on induction of anesthesia | 5 minutes prior and 15 minutes after induction of anesthesia
  The difference between the highest value before induction of anesthesia and the lowest value after induction of anesthesia will be reported.
Change of systolic blood pressure on induction of anesthesia | 5 minutes prior and 15 minutes after induction of anesthesia
  The difference between the highest value before induction of anesthesia and the lowest value after induction of anesthesia will be reported.
Change of diastolic blood pressure on induction of anesthesia | 5 minutes prior and 15 minutes after induction of anesthesia
  The difference between the highest value before induction of anesthesia and the lowest value after induction of anesthesia will be reported.
Change of mean arterial pressure on induction of anesthesia | 5 minutes prior and 15 minutes after induction of anesthesia
  The difference between the highest value before induction of anesthesia and the lowest value after induction of anesthesia will be reported.
Vasopressor | Within 15 minutes after induction of anesthesia
  Use of Vasopressors
Blood glucose level | At induction of anesthesia (Values assessed within 15 minutes prior and 15 minutes after induction of anesthesia will be accepted)
  Blood glucose level
Intravenous catheter placement | Between admission to the operation room and induction of anesthesia
  Number of attempts for placing a (first) peripheral intravenous catheter (only applicable if a peripheral intravenous catheter needs to be placed)
Postoperative nausea and vomiting | 2 hours after end of surgery
  Postoperative nausea and vomiting is a composite endpoint of the following dimensions: Vomiting, retching, nausea, and/or use of rescue medication.
Unplanned ICU/IMC | From end of surgery until last Follow-up is concluded at up to 48 hours post surgery
  Unplanned intensive/intermediate care unit stay due to respiratory complications
Number of Participants with confirmed bronchopulmonary aspiration | From induction of anesthesia until last Follow-up is concluded at up to 48 hours post surgery
  If relevant bronchopulmonary aspiration is suspected, it needs to be confirmed by bronchoscopy or radiology imaging up to 48 hours after anaesthesia procedure
All cause mortality | From end of surgery until last Follow-up is concluded at up to 48 hours post surgery
  Death within observation period
Patient satisfaction | 2 hours after end of surgery
  Patient satisfaction, operationalized using the Bauer Satisfaction Questionnaire, includes 10 ordinal items with 3 levels (where higher values indicate unfavourable outcomes), 5 items on a Likert scale with 4 levels (where lower values indicate unfavourable outcomes), and one binary item.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Meybohm, Prof. Dr., Study Director — University Hospital Würzburg, Department of Anaesthesiology, Intensive Care, Emergency and Pain Medicine, Oberdürrbacher Str. 6, 97080 Würzburg, Germany; Tobias E Haas, Dr., Principal Investigator — University Hospital Würzburg, Department of Anaesthesiology, Intensive Care, Emergency and Pain Medicine, Oberdürrbacher Str. 6, 97080 Würzburg, Germany
Locations (1):
- Wuerzburg University Hospital, Würzburg, Bavaria, Germany

REFERENCES:
- [Derived] Haas TE, Kranke P, Stegemann MN, Helmer P, Schmid B, Diehl FM, Heuschmann PU, Rucker V, Seitz AK, Diessner J, Heintel T, Saller T, Ruggeberg A, Kronert S, von Keitz J, Meybohm P. Benefits in adults allowed to drink clear liquids before anaesthesia until called to the operating room: A randomised pilot study. Eur J Anaesthesiol. 2025 Nov 19. doi: 10.1097/EJA.0000000000002309. Online ahead of print. PMID 41257406

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT06253052/Prot_SAP_000.pdf